CLINICAL TRIAL: NCT01236248
Title: Drug Abuse Prevention Among Girls Through a Mother-Daughter Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAB2130; R01DA017721 (NIH)
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Substance Use
Keywords: drugs; youth; parent; computer; prevention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevention Program (Experimental): Girls and their mothers who are assigned to participate in a tobacco, alcohol, and other drug use prevention program aimed at young girls.
  Interventions: Behavioral: Prevention
- No Prevention Program (No Intervention): Girls and their mothers who are assigned to participate in questionnaires only.

INTERVENTIONS:
Behavioral: Prevention — 9-session computerized cognitive behavioral program that young girls and their mothers interact with on a weekly basis in the privacy of their home. Girls and their mothers will watch and interact with 10 compact disc (CD) intervention sessions to learn skills to help girls avoid substance use.
  Arms: Prevention Program

SUMMARY:
The purpose of this study is to determine a computer- and family-based drug abuse prevention program is able to reduce drug use among early adolescent girls.

DETAILED DESCRIPTION:
This study longitudinally tested a computerized, parent-involvement substance abuse prevention program for adolescent girls and their mothers. The prevention program aimed to strengthen and sustain the mother-daughter bond while equipping girls with the necessary information and skills to increase protective factors and reduce risk factors associated with tobacco, alcohol, and other harmful substance use.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking New York City (NYC) area girls
* Ages 11 - 13 years
* Must have private access to a computer with high-speed connectivity

Exclusion Criteria:

* Non-English-speaking girls who do not live in the NYC area
* Younger than 11 or older than 13 years of age
* Those who lack of private access to a computer with high-speed connectivity

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 916 (Actual)
Dates: Start 2004-12; Primary Completion 2010-03 (Actual); Study Completion 2012-10-04 (Actual)

PRIMARY OUTCOMES:
Rate of Substance Use | Annually
  Measured 30-day alcohol, tobacco, and other illicit drug use among girls.

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Schinke, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States